CLINICAL TRIAL: NCT01527110
Title: An Open-label, Multi-centre, Single Arm Study to Evaluate the Safety and Efficacy of Intravenous Zanamivir in the Treatment of Hospitalized Patients With Confirmed Influenza Infection (NAI115215)
Brief Title: A Study of Intravenous Zanamivir in the Treatment of Hospitalized Patients With Influenza Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115215
Record Dates: First submitted 2011-12-08; First posted 2012-02-06 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2017-07

CONDITIONS: Influenza, Human
Keywords: zanamivir; Seasonal Influenza; H1N1; intravenous; neuraminidase inhibitor; Pandemic; Relenza; Influenza B virus; Influenza A virus
MeSH Terms: conditions — Influenza, Human | interventions — Zanamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravenous (IV) zanamivir 600mg twice daily (Experimental): 600mg of IV zanamivir infusion twice daily
  Interventions: Drug: Intravenous (IV) zanamivir

INTERVENTIONS:
Drug: Intravenous (IV) zanamivir — Zanamivir aqueous solution 10mg/mL, 600mg of IV zanamivir infusion twice daily for 5 days

SUMMARY:
This study will be an open-label, multi-center, single arm study to evaluate the safety and efficacy of IV zanamivir 600mg twice daily for 5 days in hospitalized subjects with laboratory confirmed influenza infection.

DETAILED DESCRIPTION:
Adult subjects and adolescent subjects (≥50 kg) with normal renal function will receive 600mg per dose. Subjects with renal impairment will receive an adjusted dose based on calculated creatinine clearance. The initial 5 day treatment course may be extended for up to 5 additional days if viral shedding is determined to be ongoing or if clinical symptoms warrant further treatment with IV zanamivir.

The study duration is approximately 28 days for subjects whose treatment duration is 5 days, and up to approximately 33 days for subjects whose treatment duration is extended to a maximum of 10 days. The study will consist of Pre-dose Baseline Assessments (Day 1), During Treatment Assessments (Days 1 to 5, and up to Day 10), and Follow-up Assessments on the following days: Post-Treatment +2, +5, +9, +16 and +23 Days. For subjects who have been discharged from hospital, the Post-Treatment +2, +5, +9 and +16 Days Assessments can be made by telephone contact.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged greater than or equal to 16 years of age; a female is eligible to enter and participate in the study if she is:

  1. of non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal); or,
  2. of child-bearing potential, has a negative pregnancy test at Baseline, and agrees to use protocol specified methods of birth control while on study.
* Subjects who have laboratory confirmed influenza as determined by a positive result in a rapid antigen test (RAT) for influenza A or influenza B, or a laboratory test for influenza including but not limited to influenza virus antigen test, virus culture or RT-PCR test.
* Presence of fever [oral temperature of >=38 deg C, rectal, tympanic of >=38.5 deg C or axilla >=37.4 deg C] at Baseline. However, this requirement is waived if the subject has a history of fever within the 48 hours prior to Baseline and has been administered any antipyretic(s) in the 48 hours prior to Baseline.
* Hospitalized subjects with symptomatic influenza as defined by ANY of the following.

  1. Moderate to severe tachypnea (respiratory rate >=24/minute) OR
  2. Moderate to severe dyspnea (unable to speak in full sentences) OR
  3. Arterial oxygen saturation <95% on room air by trans-cutaneous method, or need for any supplemental oxygenation or ventilatory support [mechanical ventilation, bi-level positive airway pressure (bipap), continuous positive airway pressure (cpap)], or increase in oxygen supplementation requirement of >=2 litres for subjects with chronic oxygen dependency. For those subjects with a history of chronic hypoxia (without supplemental oxygen), an arterial oxygen saturation of at least 3% below the patient's historical baseline oxygen saturation will satisfy this criterion OR
  4. Hemodynamic instability, defined as systolic blood pressure <90 mmHg or heart rate >100 beats per minute OR
  5. Subject who became dehydrated and need whole-body management by hospitalization.
* Onset of influenza symptoms within 6 days prior to study enrolment. Symptoms may include cough, dyspnea, sore throat, feverishness, myalgias, headache, nasal symptoms (rhinorrhea, congestion), fatigue, diarrhea, anorexia, nausea and vomiting.
* Subjects/legally acceptable representative of unconscious adults willing and able to give written informed consent to participate in the study, and subjects willing to adhere to the procedures stated in the protocol.

Exclusion Criteria:

* Subjects who, in the opinion of the investigator, are not likely to survive beyond 48 hours from Baseline.
* Subjects who are considered to require concurrent therapy with another influenza antiviral medication.
* Subjects who are known or suspected to be hypersensitive to any component of the study medications.
* Subjects who require Extra Corporeal Membrane Oxygenation (ECMO) at Baseline (enrolled subject who subsequently require ECMO may continue in the study).
* Liver toxicity criteria based on local laboratory results obtained at Baseline:

  1. ALT or AST >=3xULN and bilirubin >=2xULN
  2. ALT >=5xULN
* Underlying chronic liver disease with evidence of severe liver impairment (Child-Pugh Class C).
* History of severe cardiac disease or clinically significant arrhythmia (either on ECG or by history) which, in the opinion of the investigator or sub-investigator, will interfere with the safety of the individual subject.
* Females who are pregnant (positive urine or serum pregnancy test at Baseline) or are breastfeeding.
* QT criteria at Baseline as defined below:

  1. QTcB or QTcF >480 msec
  2. If a subject has bundle branch block then criteria is QTcB or QTcF >510 msec
* Subject has participated in any study using an investigational drug during the previous 30 days.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-01-01; Primary Completion 2013-03-01 (Actual); Study Completion 2013-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Japan (6):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Watanabe A, Yates PJ, Murayama M, Soutome T, Furukawa H. Evaluation of safety and efficacy of intravenous zanamivir in the treatment of hospitalized Japanese patients with influenza: an open-label, single-arm study. Antivir Ther. 2015;20(4):415-23. doi: 10.3851/IMP2922. Epub 2014 Dec 3. PMID 25470818
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 115215 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115215 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115215 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115215 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115215 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115215 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned on 20 male or female participants, aged 16 years or older years, across 6 centers of Japan from 11 January 2012 to 29 March 2013.
Pre-assignment Details: A total of 21 hospitalized Japanese participants with laboratory confirmed influenza were enrolled to receive intravenous (IV) zanamivir 600 milligram (mg) twice daily (BID) for 5 days. The course was extended for up to 5 additional days based on ongoing viral shedding or clinical symptoms requiring treatment.
Groups:
- Zanamivir 600 mg BID: Eligible participants >=18 years and adolescents >=50 kilogram (kg) with normal renal function were administered an initial dose of IV zanamivir is 600 mg followed by BID maintenance dose administered at a constant rate over approximately 30 minutes (min) for 5 days. The standard dosage for adolescent participants <50 kg was 12 mg/kg. The BID maintenance dose regimen began 12 hours after starting the initial dose infusion. Participants with renal impairment received an adjusted dose based on calculated creatinine clearance (CLcr) with the initial dose corresponding to a CLcr of > =80 milliliter per min (mL/min) for adults and for adolescent participants > = 50 kg (i.e. 600 mg) or to the appropriate weight-based dose corresponding to a CLcr > = 80 mL/min for adolescent participants <50 kg (i.e. 12 mg/kg). There was a delay of 24 to 48 hours after the initial dose before the BID maintenance dose regimen was initiated for participants with severe renal impairment.
Period: Overall Study
Arm/Group | Zanamivir 600 mg BID
Started | 21
Completed | 20
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Zanamivir 600 mg BID: Eligible participants >=18 years and adolescents >=50 kg with normal renal function were administered an initial dose of IV zanamivir is 600 mg followed by BID maintenance dose administered at a constant rate over approximately 30 min for 5 days. The standard dosage for adolescent participants <50 kg was 12 mg/kg. The BID maintenance dose regimen began 12 hours after starting the initial dose infusion. Participants with renal impairment received an adjusted dose based on calculated CLcr with the initial dose corresponding to a CLcr of > =80 mL/min for adults and for adolescent participants > = 50 kg (i.e. 600 mg) or to the appropriate weight-based dose corresponding to a CLcr > = 80 mL/min for adolescent participants <50 kg (i.e. 12 mg/kg). There was a delay of 24 to 48 hours after the initial dose before the BID maintenance dose regimen was initiated for participants with severe renal impairment.
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.3 (23.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE), Drug-related AE, Grade 3 and Grade 4 AE, Grade 3 and 4 Drug-related AE , AE Leading to Discontinuation of Study Drug or From Study, Serious AE (SAE), Drug-related SAE, Fatal AE and Drug-related Fatal AE
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, associated with liver injury and impaired liver function defined as alanine aminotransferase >=3 x upper limit of normal (ULN), and total bilirubin >=2 x ULN or international normalised ratio >1.5. The grading of AEs and SAE's for 3/4 (3= severe, 4= potentially life threatening ) and its classification as potentially drug-related was done based on the investigator's judgment.
Time Frame: Start of treatment (Day 1) up to follow-up (Day 33)
Population: Safety Population comprised of all participants who received at least one dose of IV zanamivir.
Measure: Count of Participants; unit: Participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Participants
  Any AE | 13
  Any drug-related AE | 3
  Any grade 3 and grade 4 AE | 2
  Any grade 3 and grade 4 drug -related AE | 1
  AE leading to discontinuation of study drug | 0
  AE leading to discontinuation from study | 1
  Any SAE | 4
  Any drug-related SAE | 1
  Any death | 1
  Any fatal AE | 1
  Any drug-related fatal AE | 0

2. Primary Outcome: Number of Participants With Clinical Chemistry Parameters of Alanine Amino Transferase (ALT), Alkaline Phosphatase (ALP), Creatine Kinase and Aspartate Amino Transferase (AST) Outside the Normal Reference Range at Any Time During Treatment
Description: The reference ranges for clinical chemistry parameters were ALT 5 to 45 international units per litre [IU/L]), ALP 100 to 325 IU/L, creatine kinase 60 to 270 IU/L and AST 10 to 40 IU/L. The baseline assessments were referred to assessments at Day 1. Assessments were done at Day 1, 3 and 5.
Time Frame: Baseline (Day 1) to Day 5
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Participants
  ALT, Baseline, high | 2
  ALT, Day 3, high | 2
  ALT, Day 5, high | 4
  ALP, Baseline, high | 2
  ALP, Day 3, high | 2
  ALP, Day 5, high | 2
  AST, Baseline, high | 6
  AST, Day 3, high | 6
  AST, Day 5, high | 5
  Creatine kinase, Baseline, high | 12
  Creatine kinase, Baseline, low | 2
  Creatine kinase, Day 3, high | 5
  Creatine kinase, Day 3, low | 1
  Creatine kinase, Day 5, high | 1
  Creatine kinase, Day 5, low | 4

3. Primary Outcome: Number of Participants With Clinical Chemistry Parameters of Creatinine, Direct Bilirubin and Total Bilirubin Outside the Normal Reference Range at Any Time During Treatment
Description: The reference ranges for clinical chemistry parameters were creatinine 41.548 - 69.836 micromole per litre (µmol/L), direct bilirubin 0 to 5.13 µmol/L and total bilirubin 3.42 to 20.52 µmol/L. The baseline assessments were referred to assessments at Day 1. Assessments were done at Day 1, 3 and 5.
Time Frame: Baseline (Day 1) to Day 5
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Participants
  Creatinine, Baseline, high | 8
  Creatinine, Baseline, low | 2
  Creatinine, Day 3, high | 2
  Creatinine, Day 3, low | 4
  Creatinine, Day 5, high | 2
  Creatinine, Day 5, low | 5
  Direct bilirubin, Baseline, high | 2
  Direct bilirubin, Baseline, low | 0
  Direct bilirubin, Day 3, high | 0
  Direct bilirubin, Day 3, low | 0
  Direct bilirubin, Day 5, high | 0
  Direct bilirubin, Day 5, low | 0
  Total bilirubin, Baseline, high | 1
  Total bilirubin, Baseline, low | 0
  Total bilirubin, Day 3, high | 0
  Total bilirubin, Day 3, low | 0
  Total bilirubin, Day 5, high | 0
  Total bilirubin, Day 5, low | 0

4. Primary Outcome: Number of Participants With Clinical Chemistry Parameters of Calcium, Carbon Dioxide Content/ Bicarbonate, Chloride, Magnesium, Potassium, Sodium and Urea/ Blood Urea Nitrogen (BUN) Outside the Normal Reference Range at Any Time During Treatment
Description: The reference ranges for clinical chemistry parameters were calcium 2.0958 to 2.5948 millimole per litre (mmol/L), carbon dioxide content/ bicarbonate 19.2 to 27.1 mmol/L, chloride 98 to 108 mmol/L, magnesium 0.7809 to 1.0275 mmol/L, potassium 3.5 to 5 mmol/L, sodium 137 to 147 mmol/L and urea/BUN 2.856 to 8.211 mmol/L. The baseline assessments were referred to assessments at Day 1. Assessments were done at Day 1, 3 and 5.
Time Frame: Baseline (Day 1) to Day 5
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Participants
  Calcium, Baseline, low | 9
  Calcium, Day 3, low | 10
  Calcium, Day 5, low | 10
  Carbon dioxide content/bicarbonate, Baseline, high | 1
  Carbon dioxide content/bicarbonate, Baseline, low | 6
  Carbon dioxide content/bicarbonate, Day 3, low | 1
  Carbon dioxide content/bicarbonate, Day 5, high | 1
  Carbon dioxide content/bicarbonate, Day 5, low | 1
  Chloride, Baseline, high | 1
  Chloride, Baseline, low | 5
  Chloride, Day 3, high | 2
  Chloride, Day 3, low | 1
  Urea/ BUN, Baseline, high | 5
  Urea/ BUN, Baseline, low | 2
  Urea/ BUN, Day 3, high | 3
  Urea/ BUN, Day 3, low | 2
  Urea/ BUN, Day 5, high | 2
  Urea/ BUN, Day 5, low | 2
  Magnesium, Baseline, low | 6
  Magnesium, Day 3, low | 2
  Magnesium, Day 5, low | 3
  Sodium, Baseline, low | 8
  Sodium, Day 3, low | 2
  Sodium, Day 5, low | 1
  Potassium, Baseline, low | 2
  Potassium, Day 3, low | 2
  Potassium, Day 5, low | 2

5. Primary Outcome: Number of Participants With Clinical Chemistry Parameters of Albumin and Total Protein Outside the Normal Reference Range at Any Time During Treatment
Description: The reference ranges for clinical chemistry parameters were albumin 38 to 53 grams per liter (g/L) and total protein 67 to 83 g/L. The baseline assessments were referred to assessments at Day 1. Assessments were done at Day 1, 3 and 5.
Time Frame: Baseline (Day 1) to Day 5
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Participants
  Albumin, Baseline, low | 10
  Albumin, Day 3, low | 12
  Albumin, Day 5, low | 12
  Total protein, Baseline, low | 15
  Total protein, Day 3, low | 17
  Total protein, Day 5, low | 17

6. Primary Outcome: Number of Participants With Hematology Parameters of Basophiles, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count, White Blood Cell(WBC) Count, Hemoglobin and Hematocrit Outside the Normal Reference Range at Any Time During Treatment
Description: The reference ranges for hematology parameters were basophils 0 to 2 percentage (%), eosinophils 0 to 8%, lymphocytes 18 to 49%, monocytes 2 to 10%, total neutrophils 40 to 75%, platelet count 140 to 340 giga cells per liter (GI/L), WBC count 3.3 to 9 GI/L, hemoglobin 135 to 175 g/L and haematocrit 0.397 to 0.524 ratio. The baseline assessments were referred to assessments at Day 1. Assessments were done at Day 1, 3, and 5.
Time Frame: Baseline (Day 1) to Day 5
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Participants
  Hemoglobin, Baseline, low | 11
  Hemoglobin, Day 3, low | 11
  Hemoglobin, Day 5, low | 10
  Hematocrit, Baseline, low | 11
  Hematocrit, Day 3, low | 10
  Hematocrit, Day 5, low | 10
  Lymphocytes, Baseline, low | 18
  Lymphocytes, Day 3, high | 2
  Lymphocytes, Day 3, low | 7
  Lymphocytes, Day 5, high | 2
  Lymphocytes, Day 5, low | 4
  Monocytes, Baseline, high | 7
  Monocytes, Baseline, low | 1
  Monocytes, Day 3, high | 8
  Monocytes, Day 5, high | 5
  Total neutrophils, Baseline, high | 14
  Total neutrophils, Day 3, high | 7
  Total neutrophils, Day 3, low | 2
  Total neutrophils, Day 5, high | 4
  Total neutrophils, Day 5, low | 2
  Platelet Count, Baseline, low | 6
  Platelet Count, Day 3, low | 5
  Platelet Count, Day 5, low | 4
  WBC count, Baseline, high | 5
  WBC count, Baseline, low | 2
  WBC count, Day 3, high | 3
  WBC count, Day 3, low | 2
  WBC count, Day 5, high | 1
  WBC count, Day 5, low | 2

7. Primary Outcome: Mean Change From Baseline in Albumin and Total Protein at the Indicated Time Points
Description: Albumin and total protein were measured at Baseline , Day 3 and Day 5 during the treatment period. The baseline assessments were referred to assessments at Day 1. Change from Baseline was calculated as the value at the indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1), Day 3 and Day 5
Population: Safety Population. The number of participants available at that particular time point were used for analysis.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 18
g/L
  Albumin, Day 3 | -3.2 (2.69)
  Albumin, Day 5 | -2.6 (3.20)
  Total protein, Day 3 | -4.1 (3.18)
  Total protein, Day 5 | -3.1 (4.84)

8. Primary Outcome: Mean Change From Baseline in ALT, ALP, Creatine Kinase and AST at the Indicated Time Points
Description: ALT, ALP, creatine kinase and AST were measured at Baseline, Day 3 and Day 5 during the treatment period. The baseline assessments were referred to assessments at Day 1. Change from Baseline was calculated as the value at the indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1), Day 3 and Day 5
Population: Safety population. The number of participants available at that particular time point were used for analysis.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 18
IU/L
  ALT, Day 3 | 0.2 (7.16)
  ALT, Day 5 | 3.1 (23.48)
  ALP, Day 3 | -37.1 (34.62)
  ALP, Day 5 | -27.9 (50.49)
  Creatine kinase, Day 3 | -44.8 (131.71)
  Creatine kinase, Day 5 | -192.7 (236.46)
  AST, Day 3 | -0.5 (11.95)
  AST, Day 5 | -0.2 (28.80)

9. Primary Outcome: Mean Change From Baseline in Creatinine, Direct Bilirubin and Total Bilirubin at the Indicated Time Points
Description: Creatinine, direct bilirubin and total bilirubin were measured at Baseline, Day 3 and Day 5 during the treatment period. The baseline assessments were referred to assessments at Day 1. Change from Baseline was calculated as the value at the indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1), Day 3 and Day 5
Population: Safety Population. The number of participants available at that particular time point were used for analysis.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 18
µmol/L
  Creatinine, Day 3 | -14.6351 (20.56740)
  Creatinine, Day 5 | -19.2024 (26.79556)
  Direct bilirubin, Day 3 | -0.950 (1.7812)
  Direct bilirubin, Day 5 | -0.475 (1.9280)
  Total bilirubin, Day 3 | -3.040 (4.1289)
  Total bilirubin, Day 5 | -1.520 (4.0589)

10. Primary Outcome: Mean Change From Baseline in Sodium, Calcium, Potassium, Chloride, Magnesium, Carbon Dioxide Content/Bicarbonate and Urea/BUN at the Indicated Time Points
Description: Calcium, potassium, chloride, magnesium, carbon dioxide content/bicarbonate, sodium and urea/BUN were measured at Baseline, Day 3 and Day 5 during the treatment period. The baseline assessments were referred to assessments at Day 1. Change from Baseline was calculated as the value at the indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1), Day 3 and Day 5
Population: Safety Population. The number of participants available at that particular time point were used for analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 18
mmol/L
  Calcium, Day 3 | -0.037 (0.0942)
  Calcium, Day 5 | 0.019 (0.1163)
  Potassium, Day 3 | -0.01 (0.342)
  Potassium, Day 5 | 0.02 (0.483)
  Chloride, Day 3 | 3.6 (3.27)
  Chloride, Day 5 | 3.3 (3.44)
  Magnesium, Day 3 | 0.073 (0.0941)
  Magnesium, Day 5 | 0.039 (0.0803)
  Carbon dioxide content/bicarbonate, Day 3 | 0.54 (2.249)
  Carbon dioxide content/bicarbonate, Day 5 | 1.37 (2.557)
  Sodium, Day 3 | 2.4 (3.60)
  Sodium, Day 5 | 2.8 (3.70)
  Urea/BUN, Day 3 | 0.1388 (2.42482)
  Urea/BUN, Day 5 | -1.4280 (1.69672)

11. Primary Outcome: Mean Change From Baseline in Percentage of Basophils, Eosinophils, Lymphocytes, Monocytes and Total Neutrophils at the Indicated Time Points
Description: Percentages of basophils, eosinophils, lymphocytes, monocytes and total neutrophils were measured at Baseline, Day 3 and Day 5 during the treatment period. The baseline assessments were referred to assessments at Day 1. Change from Baseline was calculated as the value at the indicated time point minus the Baseline value.
Time Frame: Baseline, Day 3 and Day 5
Population: Safety Population. The number of participants available at that particular time point were used for analysis.
Measure: Mean (Standard Deviation); unit: Percent of blood cells
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 18
Percent of blood cells
  Basophils, Day 3 | -0.04 (0.370)
  Basophils, Day 5 | -0.08 (0.448)
  Eosinophils, Day 3 | 1.57 (2.061)
  Eosinophils, Day 5 | 2.26 (2.099)
  Lymphocytes, Day 3 | 15.26 (14.123)
  Lymphocytes, Day 5 | 18.60 (13.821)
  Monocytes, Day 3 | 0.16 (4.145)
  Monocytes, Day 5 | -0.19 (4.961)
  Total neutrophils, Day 3 | -16.95 (16.483)
  Total neutrophils, Day 5 | -20.59 (17.469)

12. Primary Outcome: Mean Change From Baseline in Counts of WBC and Platelets at the Indicated Time Points
Description: WBC and platelet counts were measured at Baseline, Day 3 and Day 5 during the treatment period. The baseline assessments were referred to assessments at Day 1. Change from Baseline was calculated as the value at the indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1), Day 3 and Day 5
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
GI/L
  Platelet count, Day 3: number analyzed (Participants) | 17
  Platelet count, Day 3 | -1.6 (15.87)
  Platelet count, Day 5: number analyzed (Participants) | 16
  Platelet count, Day 5 | 14.3 (28.75)
  WBC count, Day 3: number analyzed (Participants) | 18
  WBC count, Day 3 | -1.76 (2.780)
  WBC count, Day 5: number analyzed (Participants) | 18
  WBC count, Day 5 | -1.82 (2.560)

13. Primary Outcome: Mean Change From Baseline in Hemoglobin at the Indicated Time Points
Description: Hemoglobin was measured at Baseline, Day 3 and Day 5 during the treatment period. The baseline assessments were referred to assessments at Day 1. Change from Baseline was calculated as the value at the indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1), Day 3 and Day 5
Population: Safety Population. The number of participants available at that particular time point were used for analysis.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 18
g/L
  Day 3 | -4.9 (9.10)
  Day 5 | -3.6 (9.82)

14. Primary Outcome: Mean Change Baseline in Hematocrit at the Indicated Time Points
Description: Hematocrit was measured at Baseline, Day 3 and Day 5 during the treatment period. The baseline assessments were referred to assessments at Day 1. Change from Baseline was calculated as the value at the indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1), Day 3 and Day 5
Population: Safety Population. The number of participants available at that particular time point were used for analysis.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 18
Ratio
  Day 3 | -0.0127 (0.02849)
  Day 5 | -0.0088 (0.03347)

15. Primary Outcome: Number of Participants With Toxicity Shifts From Baseline in Clinical Chemistry Over Period
Description: The reference ranges for clinical chemistry parameters were ALT 5 to 45 IU/L, ALP 100 to 325 IU/L, creatine kinase 60 to 270 IU/L, AST 10 to 40 IU/L, creatinine 41.548 to 69.836 µmol/L, direct bilirubin 0 to 5.13 µmol/L, total bilirubin 3.42 to 20.52 µmol/L, calcium 2.0958 to 2.5948 mmol/L, CO2/ bicarbonate 19.2 to 27.1 mmol/L, chloride 98 to 108 mmol/L, magnesium 0.7809 to 1.0275 mmol/L, potassium 3.5 to 5 mmol/L, sodium 137 to 147 mmol/L and urea/ BUN 2.856 to 8.211 mmol/L. The baseline assessments were referred to assessments at Day 1. Number of participants with shifts between normal range (NR) high, within NR and NR low values in hematology parameters from baseline (Day 1) at Day 3 and Day 5 is reported.
Time Frame: Baseline (Day 1), Day 3 and Day 5
Population: Safety Population. The number of participants available at that particular time point were used for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 18
Participants
  Albumin, Day 3, within NR to NR low | 5
  Albumin, Day 5, within NR to NR low | 5
  AST, Day 3, within NR to NR high | 2
  AST, Day 5, within NR to NR high | 3
  Calcium, Day 3, within NR to NR low | 4
  Calcium, Day 5, within NR to NR low | 4
  Creatine Kinase, Day 3, within NR to NR low | 1
  Creatine Kinase, Day 5, NR high to NR low | 1
  Creatine Kinase, Day 5, within NR to NR low | 2
  Chloride, Day 3, within NR to NR low | 1
  CO2 content/Bicarbonate,Day 5,within NR to NR high | 1
  Creatinine, Day 3, within NR to NR low | 3
  Creatinine, Day 5, NR high to NR low | 2
  Creatinine, Day 5, within NR to NR low | 2
  Potassium, Day 3, within NR to NR low | 1
  Potassium, Day 5, within NR to NR low | 1
  Magnesium, Day 3, within NR to NR low | 1
  Total Protein, Day 3, within NR to NR low | 5
  Total Protein, Day 5, within NR to NR low | 4
  Urea/BUN, Day 3, within NR to NR low | 1
  Urea/BUN, Day 5, within NR to NR low | 1

16. Primary Outcome: Number of Participants With Toxicity Shifts From Baseline in Hematology Parameters Over Period
Description: The reference ranges for hematology parameters were basophils 0 to 2%, eosinophils 0 to 8%, lymphocytes 18 to 49%, monocytes 2 to 10%, total neutrophils 40 to 75%, platelet count 140 to 340 GI/L, WBC count 3.3 to 9 GI/L, hemoglobin 135 to 175 g/L and haematocrit 0.397 to 0.524 ratio. The baseline assessments were referred to assessments at Day 1. Number of participants with shifts between NR high, within NR and NR low values in hematology parameters from baseline (Day 1) at Day 3 and Day 5 is reported.
Time Frame: Baseline (Day 1), Day 3 and Day 5
Population: Safety Population. The number of participants available at that particular time point were used for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 18
Participants
  Hemoglobin, Day 3, within NR to NR low | 3
  Hemoglobin, Day 5, within NR to NR low | 3
  Hematocrit, Day 3, within NR to NR low | 2
  Hematocrit, Day 5, within NR to NR low | 3
  Lymphocytes, Day 3, NR low to NR high | 2
  Lymphocytes, Day 5, NR low to NR high | 2
  Monocytes, Day 3, within NR to NR high | 3
  Monocytes, Day 3, within NR to NR low | 1
  Monocytes, Day 5, within NR to NR high | 2
  Monocytes, Day 5, within NR to NR low | 1
  Total Neutrophils, Day 3, NR high to NR low | 1
  Total Neutrophils, Day 3, within NR to NR low | 1
  Total Neutrophils, Day 5, NR high to NR low | 2
  WBC count, Day 3, within NR to NR high | 1
  WBC count, Day 3, within NR to NR low | 2
  WBC count, Day 5, within NR to NR low | 2

17. Primary Outcome: Number of Participants of Treatment Emergent Toxicities in Clinical Chemistry and Hematology Over Period
Description: The normal reference ranges for clinical chemistry and hematology parameters were ALT 5 to 45 IU/L, ALP 100 to 325 IU/L, creatine kinase 60 to 270 IU/L, AST 10 to 40 IU/L, creatinine 41.548 to 69.836 µmol/L, direct bilirubin 0 to 5.13 µmol/L, total bilirubin 3.42 to 20.52 µmol/L, calcium 2.0958 to 2.5948 mmol/L, CO2/ bicarbonate 19.2 to 27.1 mmol/L, chloride 98 to 108 mmol/L, magnesium 0.7809 to 1.0275 mmol/L, potassium 3.5 to 5 mmol/L, sodium 137 to 147 mmol/L, urea/ BUN 2.856 to 8.211 mmol/L, basophils 0 to 2%, eosinophils 0 to 8%, lymphocytes 18 to 49%, monocytes 2 to 10%, total neutrophils 40 to 75%, platelet count 140 to 340 GI/L, WBC count 3.3 to 9 GI/L, hemoglobin 135 to 175 g/L and haematocrit 0.397 to 0.524 ratio. Participants with treatment emergent toxicities for grade 3 (severe) and grade 4 (potentially life threatening) were assessed at Day 1, Day 3 and Day 5. Classification of the toxicities as potentially drug-related was done based on the investigator's judgment.
Time Frame: Day 1, Day 3 and Day 5
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Participants
  Hemoglobin decrease | 1
  Hypokalaemia | 1

18. Primary Outcome: Mean Heart Rate (HR) of Participants Over Period
Description: Vital sign of HR was assessed three times daily during the treatment period/hospitalization at Day 1, Day 2, Day 3, Day 4, Day 5 and Day 6. The baseline assessments were referred to assessments at Day 1. Maximum value in a day is reported where a 'day' is defined as a 24 h period (Treatment Day).
Time Frame: Baeline (Day 1) to Day 6
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Beats/min
  Baseline (Day 1) | 84.4 (18.76)
  Day 2 | 86.3 (19.70)
  Day 3: number analyzed (Participants) | 18
  Day 3 | 80.3 (15.88)
  Day 4: number analyzed (Participants) | 18
  Day 4 | 77.3 (13.35)
  Day 5: number analyzed (Participants) | 18
  Day 5 | 73.2 (10.96)
  Day 6: number analyzed (Participants) | 11
  Day 6 | 80.3 (10.20)

19. Primary Outcome: Mean Systolic and Diastolic Blood Pressure (SBP and DBP) of Participants Over Period
Description: Vital signs of SBP and DBP were assessed three times daily during the treatment period/hospitalization at Day 1, Day 2, Day 3, Day 4, Day 5 and Day 6. The baseline assessments were referred to assessments at Day 1. Minimum value in a day for SBP is reported where a 'day' is defined as a 24 h period (Treatment Day). DBP is measured at the same time as minimum SBP.
Time Frame: Baseline (Day 1) to Day 6
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Millimeter of mercury (mmHg)
  SBP, Baseline (Day 1) | 122.5 (20.38)
  SBP, Day 2 | 106.3 (18.49)
  SBP, Day 3: number analyzed (Participants) | 18
  SBP, Day 3 | 110.7 (17.74)
  SBP, Day 4: number analyzed (Participants) | 18
  SBP, Day 4 | 114.2 (24.42)
  SBP, Day 5: number analyzed (Participants) | 18
  SBP, Day 5 | 116.1 (18.95)
  SBP, Day 6: number analyzed (Participants) | 11
  SBP, Day 6 | 117.8 (20.13)
  DBP, Baseline (Day 1) | 71.0 (12.61)
  DBP, Day 2 | 59.0 (8.95)
  DBP, Day 3: number analyzed (Participants) | 18
  DBP, Day 3 | 63.9 (11.61)
  DBP, Day 4: number analyzed (Participants) | 18
  DBP, Day 4 | 65.2 (13.91)
  DBP, Day 5: number analyzed (Participants) | 18
  DBP, Day 5 | 66.2 (12.54)
  DBP, Day 6: number analyzed (Participants) | 11
  DBP, Day 6 | 70.5 (16.19)

20. Primary Outcome: Mean Oxygen Saturation (OS) of Participants Over Period
Description: Vital signs of OS was assessed three times daily during the treatment period/hospitalization at Day 1, Day 2, Day 3, Day 4, Day 5 and Day 6. The baseline assessments were referred to assessments at Day 1. Minimum value in a day is reported, where a 'day' is defined as a 24 h period (Treatment Day).
Time Frame: Baseline (Day 1) to Day 6
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent oxygen saturation
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Percent oxygen saturation
  Baseline (Day 1) | 95.6 (2.87)
  Day 2 | 94.1 (3.61)
  Day 3: number analyzed (Participants) | 18
  Day 3 | 95.0 (3.05)
  Day 4: number analyzed (Participants) | 18
  Day 4 | 94.2 (2.96)
  Day 5: number analyzed (Participants) | 18
  Day 5 | 94.8 (2.71)
  Day 6: number analyzed (Participants) | 11
  Day 6 | 94.6 (4.76)

21. Primary Outcome: Mean Respiratory Rate (RR) of Participants Over Period
Description: Vital signs of RR was assessed three times daily during the treatment period/hospitalization at Day 1, Day 2, Day 3, Day 4, Day 5 and Day 6. The baseline assessments were referred to assessments at Day 1. Maximum value in a day is reported, where a 'day' was defined as a 24 h period (Treatment Day).
Time Frame: Baseline (Day 1) to Day 6
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths/min
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Breaths/min
  Baseline (Day 1) | 22.9 (6.50)
  Day 2 | 22.3 (5.15)
  Day 3: number analyzed (Participants) | 18
  Day 3 | 21.7 (4.73)
  Day 4: number analyzed (Participants) | 18
  Day 4 | 21.4 (5.27)
  Day 5: number analyzed (Participants) | 18
  Day 5 | 21.2 (5.25)
  Day 6: number analyzed (Participants) | 11
  Day 6 | 21.1 (5.96)

22. Primary Outcome: Mean Temperature of Participants Over Period
Description: Vital signs of temperature was assessed three times daily during the treatment period/hospitalization at Day 1, Day 2, Day 3, Day 4, Day 5 and Day 6. The baseline assessments were referred to assessments at Day 1. Maximum value in a day is reported, where a'day' was defined as a 24 h period (Treatment Day).
Time Frame: Baseline (Day 1) to Day 6
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degrees celcius (C)
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Degrees celcius (C)
  Baseline (Day 1) | 37.75 (0.908)
  Day 2 | 37.54 (0.688)
  Day 3: number analyzed (Participants) | 18
  Day 3 | 37.01 (0.591)
  Day 4: number analyzed (Participants) | 18
  Day 4 | 36.77 (0.451)
  Day 5: number analyzed (Participants) | 8
  Day 5 | 36.67 (0.457)
  Day 6: number analyzed (Participants) | 11
  Day 6 | 36.81 (0.556)

23. Primary Outcome: Number of Participants With Abnormal Clinically Significant Electrocardiograph (ECG) Findings Over Period
Description: 12-lead ECG assessments were obtained at Baseline (Day 1) and Day 4 of the treatment period. On Baseline (Day 1), 2 baseline ECGs were obtained prior to study drug infusion. On Day 4, 2 ECGs were obtained, 1 ECG just prior to study drug infusion and 1 ECG at the end of infusion. Overall ECG findings were summarized with regard to visits at Day 1 (pre-dose [ECG 1 and ECG 2]) and Day 4 (pre-dose and 30-min post dose).
Time Frame: Baseline (Day 1, pre-dose) and Day 4
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Participants
  Baseline (Day 1), pre-dose, ECG 1 | 1
  Baseline (Day 1), pre-dose, ECG 2 | 1
  Day 4, pre-dose: number analyzed (Participants) | 18
  Day 4, pre-dose | 1
  Day 4, 30 min post-dose: number analyzed (Participants) | 18
  Day 4, 30 min post-dose | 1

24. Primary Outcome: Percentage of Participants With Abnormal Clinically Significant ECG Findings Over Period
Description: 12-lead ECG assessments were obtained at Baseline (Day 1) and Day 4 of the treatment period. On Baseline (Day 1), 2 baseline ECGs were obtained. On Day 4, 2 ECGs were obtained, 1 ECG just prior to study drug infusion and 1 ECG at the end of infusion. Overall ECG findings were summarized at Day 1 (ECG 1 and ECG 2) and Day 4 (pre-dose and 30-min post dose).
Time Frame: Baseline ( pre-dose Day 1) and Day 4
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: % of participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
% of participants
  Baseline (Day 1), pre-dose, ECG 1 | 5
  Baseline (Day 1), pre-dose, ECG 2 | 5
  Day 4, pre-dose: number analyzed (Participants) | 18
  Day 4, pre-dose | 6
  Day 4, 30 min post-dose: number analyzed (Participants) | 18
  Day 4, 30 min post-dose | 6

25. Secondary Outcome: Median Time to Absence of Fever, Improved Respiratory Status, Improved OS, Improved HR and Improved SBP Over Period
Description: Absence of fever, improved respiratory status, OS, HR and SBP was defined according to clinical response criteria as: temperature, <= 36.6 degree C-axilla or <= 37.2 degree C-oral or <= 37.7 degree C-rectal and tympanic, without the use of antipyretics within 8 hour; OS of >= 95%; respiratory status of return to pre-morbid oxygen requirement (participants with chronic oxygen use) or need for supplemental oxygen (administered by any modality) to no need for supplemental oxygen or RR <=24 breaths/min without supplemental oxygen; HR <=100 beats/min; SBP of >=90 mmHg without inotropic support within 8 hour. For OS, participants with a history of chronic hypoxia (without supplemental oxygen) satisfied normalization criteria for OS if the value without supplemental oxygen was <=2% from participants historical OS and waiver for participants with a history of chronic supplemental oxygen requirement with baseline OS <95% with supplemental oxygen, recorded within 12 months prior to enrolment.
Time Frame: Baseline (Day 1) to Day 33 (follow-up)
Population: Intent-to-Treat Exposed (ITT-E) Population comprised of all participants who receive at least one dose of IV zanamivir. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: hour
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
hour
  Absence of fever | 24.900 [9.50 to 82.33]
  Improved respiratory status: number analyzed (Participants) | 10
  Improved respiratory status | 35.140 [3.83 to 331.77]
  Improved OS: number analyzed (Participants) | 5
  Improved OS | 11.170 [3.00 to 49.60]
  Improved HR: number analyzed (Participants) | 7
  Improved HR | 6.630 [2.50 to 24.00]
  Improved SBP: number analyzed (Participants) | 4
  Improved SBP | 11.865 [2.97 to 16.50]

26. Secondary Outcome: Median Time to Clinical Response Over Period
Description: Clinical response was defined as resolution of at least 4 of the 5 vital signs within the respective resolution criteria of temperature <= 36.6 degree C-axilla or <= 37.2 degree C-oral or <= 37.7 degree C-rectal/ tympanic, without the use of antipyretics within 8 hour; OS of >= 95%; respiratory status of return to pre-morbid oxygen requirement (participants with chronic oxygen use) or need for supplemental oxygen (administered by any modality) to no need for supplemental oxygen or RR <= 24 breaths/min without supplemental oxygen; HR <=100 beats/min; SBP of >= 90 mmHg without inotropic support within 8 h, maintained for at least 24 hour, or hospital discharge, which ever occurred first. Participants discharged from hospital due to clinical improvement/resolution were considered to have met the clinical response endpoint at the time of hospital discharge and were not required to have documented resolution of at least 4 response criteria i.e. achieved success at the time of discharge.
Time Frame: Baseline (Day 1) to Day 33 (follow-up)
Population: ITT-E Population. The number of participants available at that particular time point were used for analysis.
Measure: Median (Full Range); unit: hour
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 20
hour | 85.050 [12.67 to 530.37]

27. Secondary Outcome: Median Time to Return to Pre-morbid Level of Activity Over Period
Description: Pre-morbid functional status was defined as the best functional status in the 4 weeks prior to enrolment and status at Baseline (Day 1). The participants were assessed on a 3-point scale by activity level (bed rest, limited ambulation or unrestricted) recorded in thee electronic case report form (eCRF). For participants who were unable to communicate their pre-morbid functional status, the information was requested from another close member of the household or close family member.
Time Frame: Baseline (Day 1) to Day 33 (follow-up)
Population: ITT-E Population. The number of participants available at that particular time point were used for analysis.
Measure: Median (Full Range); unit: hour
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 16
hour | 87.645 [21.00 to 714.62]

28. Secondary Outcome: Number of Participants With and Without Use of Modality of Invasive, Non-invasive Ventilatory Support and Oxygen Supplementation Over Period
Description: The non-invasive ventilator support includes modalities of machine-assisted: continuous positive airway pressure (CPAP) and bi-level positive airway pressure (BiPAP). The invasive ventilator support included modalities of machine-assisted: extra corporeal membrane oxygenation (ECMO) and endotracheal mechanical ventilation. Participants with and without use of modality of invasive, non-invasive ventilatory support and oxygen supplementation was assessed from Baseline (Day 1) to Day 33 (follow-up).
Time Frame: Baseline (Day 1) to Day 33 (follow-up)
Population: ITT-E Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Participants
  Invasive and non-invasive ventilatory support, no | 18
  Invasive and non-invasive ventilatory support, yes | 3
  CPAP | 1
  BiPAP | 1
  ECMO | 0
  Endotracheal mechanical ventilation | 2
  Oxygen supplementation, no | 10
  Oxygen supplementation, yes | 11

29. Secondary Outcome: Median Duration of Use of Invasive and Non-invasive Ventilatory Support and Oxygen Supplementation Over Period
Description: The non-invasive ventilator support includes modalities of machine-assisted: CPAP and BiPAP. The invasive ventilator support included modalities of machine-assisted: ECMO and endotracheal mechanical ventilation. Participants with use of modality of invasive, non-invasive ventilatory support and oxygen supplementation was assessed from Baseline (Day 1) to Day 33 (follow-up).
Time Frame: Baseline (Day 1) to Day 33 (follow-up)
Population: ITT-E Population. The number of participants with use of modality of invasive and non-invasive ventilatory support (3) and oxygen supplementation (11) were analysed.
Measure: Median (Full Range); unit: hour
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
hour
  Invasive and non-invasive ventilatory support: number analyzed (Participants) | 3
  Invasive and non-invasive ventilatory support | 62.330 [17.35 to 109.08]
  Oxygen supplementation: number analyzed (Participants) | 11
  Oxygen supplementation | 46.250 [0.00 to 238.75]

30. Secondary Outcome: Median Duration of Intensive Care Unit (ICU) Stay for the Participants Over Period
Description: The duration of ICU stay was assessed from the first day of dosing (Day 1) up to Day 33 (follow-up). Duration in ICU was captured from the eCRF. If the duration in ICU was missing, then the data was set to 0.
Time Frame: Baseline (Day 1) to Day 33 (follow-up)
Population: ITT-E Population.
Measure: Median (Full Range); unit: Days
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Days | 0.0 [0 to 0]

31. Secondary Outcome: Median Duration of Hospital Stay for the Participants Over Period
Description: The duration of hospital stay was assessed from the first day of dosing (Day 1) up to Day 33 (follow-up). The duration was calculated as duration in hospital = date/time of discharge - date/time of 1st day of dosing.
Time Frame: Baseline (Day 1) to Day 33 (follow-up)
Population: ITT-E Population. The number of participants available at that particular time point were used for analysis.
Measure: Median (Full Range); unit: hour
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 20
hour | 138.215 [65.17 to 530.37]

32. Secondary Outcome: Mean 50% Inhibitory Concentration (IC50) for Phenotypes of Influenza for the Measure of Viral Susceptibility to Zanamivir at All Visits
Description: IC50 value is defined as the concentration of zanamivir required to achieve half maximal inhibition of the influenza viral enzyme neuraminidase of influenza A and B to prevent the release and spread of influenza virus in the respiratory tract. Susceptibility analyses were performed on nasopharyngeal swabs collected on Baseline (Day 1) up to Day 33 (follow-up) depending on the extend of continuation of treatment and duration of hospitalization. Endotracheal aspirates were used in participants who were intubated. Data is categorized for participants with influenza A/H3N2 and influenza B.
Time Frame: Baseline (Day 1) to Day 33 (follow-up)
Population: ITT-E Population. The number of participants available at that particular time point were used for analysis.
Measure: Mean (Standard Deviation); unit: Nanomole per liter (nmol/L)
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 18
Nanomole per liter (nmol/L)
  Influenzavirus A/H3N2, at all visits: number analyzed (Participants) | 15
  Influenzavirus A/H3N2, at all visits | 2.04 (0.275)
  Influenzavirus B, at all visits: number analyzed (Participants) | 3
  Influenzavirus B, at all visits | 8.85 (1.277)

33. Secondary Outcome: Number of Participants With or Without Treatment Emergent Resistance or Suspected Treatment Emergent Resistance to Zanamivir Over Period
Description: A total of 30 neuraminidase gene sequences (23 influenza A/H3N2, 5 influenza B and 2 negative) from 21 participants were obtained from 76 samples. There were no resistance associated neuraminidase mutations or mutations in the neuraminidase active site identified in viruses isolated during this study. Therefore the frequency of resistance emergence to zanamivir could not be determined.
Time Frame: Baseline (Day 1) to Day 33 (follow-up)
Population: ITT-E Population. The number of participants with Influenza A/H3N2 (17) and Influenzavirus B (3) were used for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 20
Participants
  Influenza A/H3N2, resistence or suspected: number analyzed (Participants) | 17
  Influenza A/H3N2, resistence or suspected | 0
  Influenza A/H3N2, without resistence: number analyzed (Participants) | 17
  Influenza A/H3N2, without resistence | 17
  Influenzavirus B, resistence or suspected: number analyzed (Participants) | 3
  Influenzavirus B, resistence or suspected | 0
  Influenzavirus B, without resistence: number analyzed (Participants) | 3
  Influenzavirus B, without resistence | 3

34. Secondary Outcome: Number of Participants of Clinical Symptoms of Influenza Over Period
Description: Influenza symptoms were assessed at Baseline (pre-dose): the presence of the following symptoms were recorded: nasal symptoms (rhinorrhea, congestion), feverishness, cough, myalgias, fatigue, diarrhea, anorexia, dyspnea, headache, sore throat, nausea and vomiting. The investigator assessed and recorded influenza symptoms based on interview with the participants. In cases where participants were not able to communicate their symptoms, in participants ventilated and/or sedated, the investigator recorded those signs/symptoms as 'unable to assess'.
Time Frame: Baseline (Day 1) to Day 33 (follow-up)
Population: ITT-E Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Participants
  Cough | 20
  Dyspnea | 15
  Nausea | 2
  Diarrhea | 6
  Feverishness | 19
  Fatigue | 16
  Sore throat | 7
  Headache | 10
  Nasal symptoms | 13
  Myalgias | 8
  Anorexia | 15

35. Secondary Outcome: Median Duration of Clinical Symptoms of Influenza Over Period
Description: Influenza symptoms were assessed at Baseline (pre-dose) and throughout the study period as presence of the following symptoms were recorded: nasal symptoms (rhinorrhea, congestion), feverishness, cough, myalgias, fatigue, diarrhea, anorexia, dyspnea, headache, sore throat, nausea and vomiting. The investigator assessed and recorded influenza symptoms based on interview with the participants. In cases where participants were not able to communicate their symptoms, in participants ventilated and/or sedated, the investigator recorded those signs/symptoms as 'unable to assess'.
Time Frame: Baseline (Day 1) to Day 33 (follow-up)
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Days
  Cough: number analyzed (Participants) | 20
  Cough | 7.0 [1 to 25]
  Dyspnea: number analyzed (Participants) | 15
  Dyspnea | 1.0 [1 to 3]
  Nausea and vomiting: number analyzed (Participants) | 2
  Nausea and vomiting | 1.0 [1 to 1]
  Diarrhea: number analyzed (Participants) | 6
  Diarrhea | 2.0 [1 to 23]
  Feverishness: number analyzed (Participants) | 19
  Feverishness | 3.0 [1 to 30]
  Fatigue: number analyzed (Participants) | 16
  Fatigue | 3.0 [1 to 11]
  Sore throat: number analyzed (Participants) | 7
  Sore throat | 2.0 [1 to 3]
  Headache: number analyzed (Participants) | 10
  Headache | 1.5 [1 to 3]
  Nasal symptoms: number analyzed (Participants) | 13
  Nasal symptoms | 2.0 [1 to 30]
  Myalgias: number analyzed (Participants) | 8
  Myalgias | 2.0 [1 to 3]
  Anorexia: number analyzed (Participants) | 15
  Anorexia | 2.0 [1 to 8]

36. Secondary Outcome: Number of Participants With Complications of Influenza and Associated Use of Antibiotics Over Period
Description: The details of complications of influenza like bacterial pneumonia, pneumothorax, pleural effusion, acute respiratory distress syndrome (ARDS), myositis, encephalitis, myocarditis and associated antibiotic use were assessed from Baseline (Day 1) to Day 33 (follow-up). Participants with complications of influenza, with associated use of antibiotics as " associated antibiotic use yes" and without associated use of antibiotics as "associated antibiotic use no" were categorized.
Time Frame: Baseline (Day 1) to Day 33 (follow-up)
Population: ITT-E Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Participants
  Complications of influenza | 11
  Associated antibiotic use, no | 0
  Associated antibiotic use, yes | 11

37. Secondary Outcome: Median Time to Virologic Improvement Over Period
Description: Virologic improvement was defined as a 2 log drop in viral load or sustained undetectable viral ribonucleic acid (RNA), on 2 successive occasions as measured by quantitative reverse transcriptase - polymerase chain reaction (RT-PCR) from nasopharyngeal samples. Assessment was done from Baseline (Day 1) up to Day 33 (follow-up).
Time Frame: Baseline (Day 1) to Day 33 (follow-up)
Population: ITT-E Population. The number of participants available at that particular time point were used for analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 19
Days | 3.0 [2 to 5]

38. Secondary Outcome: Percentage of Participants With Undetectable Viral RNA and Absence Cultivable Virus From Samples Obtained From Nasopharyngeal Samples Over Period
Description: Quantitative RT-PCR and quantitative viral culture was carried out on nasopharyngeal swabs collected from Baseline (Day 1) up to Day 33 (follow-up) depending on the extend of continuation of treatment and duration of hospitalization of the participants. Undetectable RNA concentrations were below the level of quantification.
Time Frame: Baseline (Day 1) to Day 33 (follow-up)
Population: ITT-E Population.
Measure: Number; unit: % of participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
% of participants
  BASELINE (DAY 1) | 5
  DAY 2 | 5
  DAY 3 | 5
  DAY 4 | 19
  DAY 5 | 19
  DAY 6 | 29
  LAST DAY | 38

39. Secondary Outcome: Percentage of Participants With Undetectable Viral RNA and Absence of Cultivable Virus in Lower Respiratory Samples Over Period
Description: Quantitative RT-PCR and quantitative viral culture was carried out on lower respiratory samples (endotracheal aspirates) collected on Baseline (Day 1) up to Day 33 (follow-up) depending on the extend of continuation of treatment and duration of hospitalization. Endotracheal aspirates were used in participants who were intubated. Undetectable RNA concentrations were below the level of quantification.
Time Frame: Baseline (Day 1) to Day 33 (follow-up)
Population: ITT-E Population.
Measure: Number; unit: % of participants
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
% of participants
  BASELINE (DAY 1) | 0
  DAY 2 | 0
  DAY 3 | 0
  DAY 4 | 0
  DAY 5 | 0

40. Secondary Outcome: Median Time to no Detectable Viral RNA by Quantitative RT-PCR and Viral Culture From Nasopharyngeal Samples Over Period
Description: Quantitative RT-PCR and quantitative viral culture was carried out on nasopharyngeal swabs collected on Baseline (Day 1) up to Day 33 (follow-up) depending on the extend of continuation of treatment and duration of hospitalization.
Time Frame: Baseline (Day 1) to Day 33 (follow-up)
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
Days
  Viral RNA by quantitative RT-PCR: number analyzed (Participants) | 10
  Viral RNA by quantitative RT-PCR | 5.5 [4 to 7]
  Quantitative viral culture: number analyzed (Participants) | 17
  Quantitative viral culture | 3.0 [2 to 4]

41. Secondary Outcome: Mean Change From Baseline in Quantitative Viral Load Measured by RT-PCR From Nasopharyngeal Swabs Positive at Baseline Over Period
Description: Quantitative RT-PCR was carried out on nasopharyngeal swabs collected on Day 1 up to Day 33 (last day) depending on the extend of continuation of treatment and duration of hospitalization. The baseline assessments were referred to assessments at Day 1. Change from Baseline was calculated as the value at the indicated time point minus the Baseline value. Analysis was done for participants with positive Influenza A RNA and Influenza B RNA. Data is presented for Day 3, Day 5 and last day.
Time Frame: Baseline (Day 1) up to Day 33 (follow-up)
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Logarithmic base 10 (log 10) copies/mL
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 20
Logarithmic base 10 (log 10) copies/mL
  Influenza A RNA, Day 3: number analyzed (Participants) | 14
  Influenza A RNA, Day 3 | -2.53 (1.683)
  Influenza A RNA, Day 5: number analyzed (Participants) | 14
  Influenza A RNA, Day 5 | -3.77 (1.759)
  Influenza A RNA, Last Day (Day 33): number analyzed (Participants) | 17
  Influenza A RNA, Last Day (Day 33) | -4.13 (1.938)
  Influenza B RNA, Day 3: number analyzed (Participants) | 3
  Influenza B RNA, Day 3 | -2.01 (1.973)
  Influenza B RNA, Day 5: number analyzed (Participants) | 3
  Influenza B RNA, Day 5 | -3.73 (1.712)
  Influenza B RNA, Last Day (Day 33): number analyzed (Participants) | 3
  Influenza B RNA, Last Day (Day 33) | -4.43 (1.630)

42. Secondary Outcome: Mean Change From Baseline in Quantitative Viral Load Measured by Viral Culture From Nasopharyngeal Swabs Over Period
Description: Quantitative viral culture as 50 % tissue culture infectious dose (TCID50) defined as median tissue culture infective dose is that amount of a pathogenic agent that produces pathological change in 50% of cell cultures inoculated. It was carried out on nasopharyngeal swabs collected on Day 1 up to Day 33 (last day) depending on the extend of continuation of treatment and duration of hospitalization. The baseline assessments were referred to assessments at Day 1. Change from Baseline was calculated as the value at the indicated time point minus the Baseline value. Any undetectable viral load values were calculated as x.x Log10 TCID50: x.x Log10 (1.5 or 7.5 was the lower or upper limit of quantification in TCID50). Data is presented for Day 3, Day 5 and last day.
Time Frame: Baseline (Day 1) up to Day 33 (follow-up)
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: LOG TCID50/mL
Arm/Group | Zanamivir 600 mg BID
Number analyzed (Participants) | 21
LOG TCID50/mL
  Day 3: number analyzed (Participants) | 17
  Day 3 | -2.10 (1.981)
  Day 5: number analyzed (Participants) | 18
  Day 5 | -2.23 (1.989)
  Last Day (Day 33) | -2.14 (1.958)

ADVERSE EVENTS:
Time Frame: Up to Day 33
Description: Safety Population was used which comprised of all participants who received at least one dose of IV zanamivir.
Arm/Group | Zanamivir 600 mg BID
All-Cause Mortality (participants affected / at risk) | 1/21
Serious Adverse Events (participants affected / at risk) | 4/21
Other Adverse Events (participants affected / at risk) | 4/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zanamivir 600 mg BID (N=21)
Pneumonia bacterial (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Hyperthyroidism (Endocrine disorders) | 1
Haemoglobin decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zanamivir 600 mg BID (N=21)
Diarrhoea (Gastrointestinal disorders) | 4
Pyrexia (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.